CLINICAL TRIAL: NCT06654466
Title: Enhancing Information Management for Young Adults After Genetic Cancer Risk Testing
Brief Title: Closing the GAPS: Guideline Adherence, Prevention and Surveillance in Hereditary Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nest Genomics (Industry)
Collaborators: Dana-Farber Cancer Institute (Other); National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-657; 1R42HG013908-01 (NIH)
Record Dates: First submitted 2024-10-18; First posted 2024-10-23 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hereditary Cancer Syndromes; Clinical Decision Support
Keywords: Hereditary Cancer Syndromes; Cancer Surveillance; Cancer Prevention; Guideline Adherence; Clinical Decision Support; Adolescent and Young Adult Cancer
MeSH Terms: conditions — Neoplastic Syndromes, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Patients in the control arm will complete a standard genetic counseling or follow-up visit and a post-visit survey.
- Intervention Arm (Experimental): Patients in the intervention arm will complete a genetic counseling or follow-up visit with a clinician using Nest Clinical Decision Support and a post visit-survey. Intervention arm patients will be given access to the Nest Patient Navigator.
  Interventions: Device: Nest, an electronic medical record (EMR)-integrated software platform to deliver longitudinal, genetics-based care at scale.

INTERVENTIONS:
Device: Nest, an electronic medical record (EMR)-integrated software platform to deliver longitudinal, genetics-based care at scale. — The Nest software platform includes the Nest Care Studio, Nest Patient Navigator and the Analytics Dashboard. Nest Care Studio is a clinician facing portal that can be used standalone or electronic medical record (EMR) integrated. Care Studio enables clinicians to effectively manage patients' genetic information over time. Clinicians can see a list of patients that meet criteria for testing, run risk assessment calculations, order genetic tests, manage patients based on results and view education modules.The Nest Patient Navigator is a secure mobile device accessible platform that provides a centralized location for patients to store, manage, and follow-up with their genetic results. The Analytics Dashboard is an interactive dashboard that can track outcomes of genomic programs and trigger interventions to optimize them.
  Arms: Intervention Arm

SUMMARY:
The goal of this clinical trial is to see if a software platform can improve cancer screening in young adults with genetic risk for cancer.

The trial will also help improve the software platform (Nest). The main questions it aims to answer are:

* Do Nest users know more about their cancer risks and recommended care than non-users?
* Do Nest users have less psychological distress than non-users?
* Do Nest users share cancer risks with family and other doctors more than non-users?
* Are Nest users more likely than non-users to have up-to-date care plans?

Researchers will compare Nest users to non-users to see if the Nest users are more likely to do recommended cancer screening.

Participants will:

* Have a genetic counseling or follow up visit
* Take a post-visit survey
* Intervention arm only: use the Nest Patient Navigator
* Complete screening and follow-up care recommended by doctors

DETAILED DESCRIPTION:
The overall objective of this project is to refine and study Nest, a software platform that integrates genetic data into patient care, with a goal of improving adherence to recommended care and empowering patients and clinicians to utilize genetic information longitudinally. Nest stores structured genetic results in the electronic medical record (EMR) and provides an interface for clinicians to order guidelines-based, personalized care plans with automated charting. For patients, the mobile friendly platform serves as a secure tool to store results, understand risks and recommended care, adhere to care, and share results with at-risk relatives. To facilitate continuity of care, patients can share genetic results and care plans with other clinicians. For this application, the investigators propose two phases. During Phase 1, the investigators will pilot the EMR-integrated Nest platform to ensure that the intervention is feasible and acceptable to clinicians and patients. Phase 2 will test Nest efficacy to improve patient and clinician experiences and outcomes, including patient knowledge of cancer risks and recommended care, and will assess implementation outcomes to facilitate future dissemination. The investigators will leverage a team with complementary expertise in genomic data, business, software development, and care of young adults with cancer risk. This team has already successfully collaborated in development of a patient-facing intervention for adolescents and young adults (AYAs) with cancer risk syndromes, and now seeks to meet the critical need for integrated and coordinated care, crossing patients, clinicians, and health systems. The long-term goal of this application is to harness an EMR integrated platform to improve care and outcomes for AYAs with cancer risk syndromes, as an initial step toward genomic data integration for an ever-increasing array of conditions with clinical implications.

Phase 1 Aims:

Aim 1: Pilot Nest among 20 young adult hereditary cancer patients and up to 20 clinicians, refining implementation to ensure feasibility and acceptability. Our working hypothesis is that the Nest intervention will be feasible and acceptable to patients and clinicians.

Phase 2 Aims:

In Phase 2, the investigators will Implement the Nest intervention by conducting a randomized trial at a single large cancer center and its associated community-based satellites.

Aim 1: Measure the impact of the Nest intervention on patient knowledge of cancer risk and recommended care, psychological distress, and information sharing with family and clinicians.

Our working hypothesis is that patients assigned to the Nest intervention will have increased knowledge of cancer risks and recommended care, without increased psychological distress, and will have increased frequency of information sharing with family and other clinicians.

Aim 2: Examine impact of the Nest intervention on clinician behavior, including guideline-concordant orders and referrals as well as EMR documentation. Our working hypothesis is that patients assigned to the Nest intervention will have higher rates of guidelines-concordant orders and referrals and Nest Clinical Decision Support (CDS) summaries in EMR documentation.

Aim 3: Evaluate implementation outcomes, including patient and clinician utilization of Nest features, to facilitate future dissemination. The investigators will examine the frequency of utilization of Nest features, including patient access and sharing of information and clinician use of orders and documentation templates, to assess features that are most useful and/or in need of further refinement.

Impact: At the completion of the proposed research, our expected outcomes are: to have a refined platform that results in increased knowledge, information sharing, and guidelines concordant care.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-49 years, inclusive
* previous cancer genetic testing with a finding of a pathogenic or likely pathogenic variant resulting in an increased risk of cancer warranting clinical management.
* English-speaking and -reading
* Receiving care at Dana Farber Cancer Institute
* Not in active cancer therapy at the time of approach

Exclusion Criteria:

* Age <18 or >49 years
* Has not had genetic testing for hereditary cancer syndromes or has been tested but no pathogenic or likely pathogenic variant was identified.
* Non-English speaking and reading
* Not receiving care at Dana Farber Cancer Institute
* Active cancer with therapy in progress

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure (AIM) | within 7 days of visit
  A 4-item measure of intervention acceptability on a 5-point Likert response scale designed for a range of stakeholders. Demonstrated to be associated with intervention success.
Gist Comprehension of Genetic Cancer Risk | Baseline, within 7 days of visit
  Modified items from the Gist Comprehension of Genetic Cancer Risk (alpha=.85) ask patients their likelihood of future cancer on a 5-point Likert scale, higher score indicating greater comprehension.
Knowledge of Cancer Screening | Baseline, within 7 days of visit
  An 11-item true-false scale (Cronbach's alpha=.81) will measure knowledge of cancer screening recommendations. Higher score indicates greater knowledge, minimum score=0, maximum score=11. Items will be modified for cancer risk syndromes under study.
Psychosocial Aspects of Hereditary Cancer (PAHC) | Baseline, within 7 days of visit
  A 26-item questionnaire organized into six problem domains: genetics, practical issues, family, living with cancer, emotions, and children. Higher score indicates greater emotional distress. Validated in adults with hereditary cancer risk.
Distress Thermometer (DT) | Baseline, within 7 days of visit
  A visual-analog scale from 0-"no distress" to 10-"extreme distress" to assess general psychological distress. Higher score indicates greater distress. Pairing with the PAHC enhances sensitivity and specificity.

SECONDARY OUTCOMES:
Uncertainty of Illness Measures | Baseline, within 7 days of visit
  self-report - Mischel Illness Uncertainty Scale (Cronbach's α=.74-.92).5-point Likert scale ranging from "Strongly Agree" to "Strongly Disagree". Higher scores indicate greater uncertainty.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Q Rana, MD, Principal Investigator — Dana-Farber Cancer Institute; Jennifer W Mack, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Nest Genomics — https://www.nestgenomics.com/